CLINICAL TRIAL: NCT01114607
Title: A Single Dose, Randomized, Five-Period Crossover Study to Assess the Relative Bioavailability of Four New Formulations of the CCR9 Receptor Antagonist GSK1605786A (CCX282) in Healthy Male and Female Subjects
Brief Title: A Study to Assess the Relative Bioavailability of Four New Formulations of GSK1605786 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 114203
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Crohn's Disease
Keywords: GSK1605786; relative bioavailability; CCR9 receptor antagonist
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- Treatment sequence ABCDE (Experimental): Eligible subjects will be randomized in sequence ABCDE and will receive: A= two capsules of GSK1605786 ChemoCentryx formulation 250 milligrams once daily, B= two capsules of GSK1605786 GSK formulation 250 milligrams once daily, C= two capsules of GSK1605786 GSK direct-fill formulation 250 milligrams once daily, D= two capsules of GSK1605786 GSK modified-process formulation 250 milligrams once daily, and E= film coated tablet of GSK1605786 GSK formulation 500 mg once daily.
  Interventions: Drug: GSK1605786 ChemoCentryx: formulation A; Drug: GSK1605786 GSK: formulation B; Drug: GSK1605786 GSK direct-fill: formulation C; Drug: GSK1605786 GSK modified-process: formulation D; Drug: GSK1605786 GSK tablet: formulation E
- Treatment sequence ABDEC (Experimental): Eligible subjects will be randomized in sequence ABDEC and will receive: A= two capsules of GSK1605786 ChemoCentryx formulation 250 milligrams once daily, B= two capsules of GSK1605786 GSK formulation 250 milligrams once daily, D= two capsules of GSK1605786 GSK modified-process formulation 250 milligrams once daily, E= film coated tablet of GSK1605786 GSK formulation 500 mg once daily, and C= two capsules of GSK1605786 GSK direct-fill formulation 250 milligrams once daily.
  Interventions: Drug: GSK1605786 ChemoCentryx: formulation A; Drug: GSK1605786 GSK: formulation B; Drug: GSK1605786 GSK direct-fill: formulation C; Drug: GSK1605786 GSK modified-process: formulation D; Drug: GSK1605786 GSK tablet: formulation E
- Treatment sequence ABECD (Experimental): Eligible subjects will be randomized in sequence ABECD and will receive: A= two capsules of GSK1605786 ChemoCentryx formulation 250 milligrams once daily, B= two capsules of GSK1605786 GSK formulation 250 milligrams once daily, E= film coated tablet of GSK1605786 GSK formulation 500 mg once daily, C= two capsules of GSK1605786 GSK direct-fill formulation 250 milligrams once daily, and D= two capsules of GSK1605786 GSK modified-process formulation 250 milligrams once daily.
  Interventions: Drug: GSK1605786 ChemoCentryx: formulation A; Drug: GSK1605786 GSK: formulation B; Drug: GSK1605786 GSK direct-fill: formulation C; Drug: GSK1605786 GSK modified-process: formulation D; Drug: GSK1605786 GSK tablet: formulation E
- Treatment sequence ABCED (Experimental): Eligible subjects will be randomized in sequence ABCED and will receive: A= two capsules of GSK1605786 ChemoCentryx formulation 250 milligrams once daily, B= two capsules of GSK1605786 GSK formulation 250 milligrams once daily, C= two capsules of GSK1605786 GSK direct-fill formulation 250 milligrams once daily, E= a film coated tablet of GSK1605786 GSK formulation 500 mg once daily and D= two capsules of GSK1605786 GSK modified-process formulation 250 milligrams once daily.
  Interventions: Drug: GSK1605786 ChemoCentryx: formulation A; Drug: GSK1605786 GSK: formulation B; Drug: GSK1605786 GSK direct-fill: formulation C; Drug: GSK1605786 GSK modified-process: formulation D; Drug: GSK1605786 GSK tablet: formulation E
- Treatment sequence ABDCE (Experimental): Eligible subjects will be randomized in sequence ABDCE and will receive: A= two capsules of GSK1605786 ChemoCentryx formulation 250 milligrams once daily, B= two capsules of GSK1605786 GSK formulation 250 milligrams once daily, D= two capsules of GSK1605786 GSK modified-process formulation 250 milligrams once daily, C= two capsules of GSK1605786 GSK direct-fill formulation 250 milligrams once daily, and E= film coated tablet of GSK1605786 GSK formulation 500 mg once daily.
  Interventions: Drug: GSK1605786 ChemoCentryx: formulation A; Drug: GSK1605786 GSK: formulation B; Drug: GSK1605786 GSK direct-fill: formulation C; Drug: GSK1605786 GSK modified-process: formulation D; Drug: GSK1605786 GSK tablet: formulation E
- Treatment sequence ABEDC (Experimental): Eligible subjects will be randomized in sequence ABEDC and will receive: A= two capsules of GSK1605786 ChemoCentryx formulation 250 milligrams once daily, B= two capsules of GSK1605786 GSK formulation 250 milligrams once daily, E= film coated tablet of GSK1605786 GSK formulation 500 mg once daily, D= two capsules of GSK1605786 GSK modified-process formulation 250 milligrams once daily, and C= two capsules of GSK1605786 GSK direct-fill formulation 250 milligrams once daily.
  Interventions: Drug: GSK1605786 ChemoCentryx: formulation A; Drug: GSK1605786 GSK: formulation B; Drug: GSK1605786 GSK direct-fill: formulation C; Drug: GSK1605786 GSK modified-process: formulation D; Drug: GSK1605786 GSK tablet: formulation E
- Treatment sequence BACDE (Experimental): Eligible subjects will be randomized in sequence BACDE and will receive: B= two capsules of GSK1605786 GSK formulation 250 milligrams once daily, A= two capsules of GSK1605786 ChemoCentryx formulation 250 milligrams once daily, C= two capsules of GSK1605786 GSK direct-fill formulation 250 milligrams once daily, D= two capsules of GSK1605786 GSK modified-process formulation 250 milligrams once daily, and E= film coated tablet of GSK1605786 GSK formulation 500 mg once daily.
  Interventions: Drug: GSK1605786 ChemoCentryx: formulation A; Drug: GSK1605786 GSK: formulation B; Drug: GSK1605786 GSK direct-fill: formulation C; Drug: GSK1605786 GSK modified-process: formulation D; Drug: GSK1605786 GSK tablet: formulation E
- Treatment sequence BADEC (Experimental): Eligible subjects will be randomized in sequence BADEC and will receive: B= two capsules of GSK1605786 GSK formulation 250 milligrams once daily, A= two capsules of GSK1605786 ChemoCentryx formulation 250 milligrams once daily, D= two capsules of GSK1605786 GSK modified-process formulation 250 milligrams once daily, E= film coated tablet of GSK1605786 GSK formulation 500 mg once daily, and C= two capsules of GSK1605786 GSK direct-fill formulation 250 milligrams once daily.
  Interventions: Drug: GSK1605786 ChemoCentryx: formulation A; Drug: GSK1605786 GSK: formulation B; Drug: GSK1605786 GSK direct-fill: formulation C; Drug: GSK1605786 GSK modified-process: formulation D; Drug: GSK1605786 GSK tablet: formulation E
- Treatment sequence BAECD (Experimental): Eligible subjects will be randomized in sequence BAECD and will receive: B= two capsules of GSK1605786 GSK formulation 250 milligrams once daily, A= two capsules of GSK1605786 ChemoCentryx formulation 250 milligrams once daily, E= film coated tablet of GSK1605786 GSK formulation 500 mg once daily, C= two capsules of GSK1605786 GSK direct-fill formulation 250 milligrams once daily, and D= two capsules of GSK1605786 GSK modified-process formulation 250 milligrams once daily.
  Interventions: Drug: GSK1605786 ChemoCentryx: formulation A; Drug: GSK1605786 GSK: formulation B; Drug: GSK1605786 GSK direct-fill: formulation C; Drug: GSK1605786 GSK modified-process: formulation D; Drug: GSK1605786 GSK tablet: formulation E
- Treatment sequence BACED (Experimental): Eligible subjects will be randomized in sequence BACED and will receive: B= two capsules of GSK1605786 GSK formulation 250 milligrams once daily, A= two capsules of GSK1605786 ChemoCentryx formulation 250 milligrams once daily, C= two capsules of GSK1605786 GSK direct-fill formulation 250 milligrams once daily, E= film coated tablet of GSK1605786 GSK formulation 500 mg once daily, and D= two capsules of GSK1605786 GSK modified-process formulation 250 milligrams once daily.
  Interventions: Drug: GSK1605786 ChemoCentryx: formulation A; Drug: GSK1605786 GSK: formulation B; Drug: GSK1605786 GSK direct-fill: formulation C; Drug: GSK1605786 GSK modified-process: formulation D; Drug: GSK1605786 GSK tablet: formulation E
- Treatment sequence BADCE (Experimental): Eligible subjects will be randomized in sequence BADCE and will receive: B= two capsules of GSK1605786 GSK formulation 250 milligrams once daily, A= two capsules of GSK1605786 ChemoCentryx formulation 250 milligrams once daily, D= two capsules of GSK1605786 GSK modified-process formulation 250 milligrams once daily, C= two capsules of GSK1605786 GSK direct-fill formulation 250 milligrams once daily, and E= film coated tablet of GSK1605786 GSK formulation 500 mg once daily.
  Interventions: Drug: GSK1605786 ChemoCentryx: formulation A; Drug: GSK1605786 GSK: formulation B; Drug: GSK1605786 GSK direct-fill: formulation C; Drug: GSK1605786 GSK modified-process: formulation D; Drug: GSK1605786 GSK tablet: formulation E
- Treatment sequence BAEDC (Experimental): Eligible subjects will be randomized in sequence BAEDC and will receive: B= two capsules of GSK1605786 GSK formulation 250 milligrams once daily, A= two capsules of GSK1605786 ChemoCentryx formulation 250 milligrams once daily, E= film coated tablet of GSK1605786 GSK formulation 500 mg once daily, D= two capsules of GSK1605786 GSK modified-process formulation 250 milligrams once daily, and C= two capsules of GSK1605786 GSK direct-fill formulation 250 milligrams once daily.
  Interventions: Drug: GSK1605786 ChemoCentryx: formulation A; Drug: GSK1605786 GSK: formulation B; Drug: GSK1605786 GSK direct-fill: formulation C; Drug: GSK1605786 GSK modified-process: formulation D; Drug: GSK1605786 GSK tablet: formulation E

INTERVENTIONS:
Drug: GSK1605786 ChemoCentryx: formulation A — ChemoCentryx formulation A will be an opaque Swedish orange body, blue coloured capsule with size zero, administered 30 minutes after standard breakfast.
Drug: GSK1605786 GSK: formulation B — GSK1605786 formulation B will be an opaque Swedish orange body capsule with size 0, administered 30 minutes after standard breakfast.
Drug: GSK1605786 GSK direct-fill: formulation C — GSK1605786 formulation C will be an opaque Swedish orange body capsule with size 1, administered 30 minutes after standard breakfast.
Drug: GSK1605786 GSK modified-process: formulation D — GSK1605786 formulation D will be an opaque Swedish orange body capsule with size 0, administered 30 minutes after standard breakfast.
Drug: GSK1605786 GSK tablet: formulation E — GSK1605786 formulation D will be a pink coloured film coated tablet, administered 30 minutes after standard breakfast.

SUMMARY:
This is an open-label, single dose, randomized, five-period, crossover study in healthy volunteers to assess the relative bioavailability of four GSK developed oral formulations of GSK1605786 relative to the capsule formulation administered in the ChemoCentryx Phase IIb, PROTECT-1 Study and ChemoCentryx Thorough QT/QTc Study.

Approximately 24 subjects will be randomized to receive a single 500 mg dose of each of the five formulations of GSK1605786 after a standard breakfast. Serial pharmacokinetic samples will be collected following each dose and safety assessments will be performed. The relative bioavailability of the GSK capsule formulation will be compared to the ChemoCentryx formulation while the relative bioavailability the three other formulations will be compared to the GSK capsule formulation intended for use in a GlaxoSmithKline Phase IIb study.

DETAILED DESCRIPTION:
This will be a randomized, open-label, single-dose, five-period, crossover study in healthy volunteers to compare the relative bioavailability of 5 oral GSK1605786 formulations. Recruitment/screening will occur within approximately 30 days of the first scheduled dose of study medication. Each subject will participate in five dosing sessions - each dose will be separated by at least seven days. The total duration of a subject's participation in the study, from Screening to Follow-up, is approximately 10 weeks.

All subjects will receive single 500mg doses of the following five GSK1605786 formulations: A. ChemoCentryx formulation of GSK1605786; 2 x 250mg capsules [Formulation A] B. GSK formulation of GSK1605786; 2 x 250mg capsules [Formulation B] C. GSK direct-fill formulation of GSK1605786; 2 x 250mg capsules [Formulation C] D. GSK modified formulation of GSK1605786; 2 x 250mg capsules [Formulation D] E. GSK tablet formulation of GSK1605786; 500mg tablet [Formulation E]

Formulations A and B will administered in periods 1 and 2 in a random order, and formulations C, D and E will be administered in periods 3, 4, and 5 in a random order.

Subjects will check into the clinical research unit (CRU) 1 day prior to dosing (Day -1). The study medication will be administered in the morning of Day 1 with 240 mL of water 30 minutes after a standard breakfast (i.e., fed state). For each treatment period, subjects will stay in the CRU through the 48-hour PK sample on the morning of Day 3. Subjects may be released from the clinic on Day 3 (after all required study procedures are completed) and return to the CRU that evening and the next morning for collection of the 60- and 72-hour PK samples.

Upon completion of the last dosing period or early withdrawal, subjects will return to the clinic approximately seven days after the last dose of study medication for a follow up visit and be subsequently discharged from the study.

The study will be conducted at one center.

ELIGIBILITY:
Inclusion Criteria:

1. AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
2. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
3. Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
4. A female subject is eligible to participate if she is of:

   * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
   * Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 4 weeks post-last dose.
5. Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 4 weeks post-last dose.
6. Body weight ≥ 50 kg (110lbs) for men and ≥45 kg (99 lbs) for women, and BMI within the range 18.5 - 31 kg/m2 (inclusive).
7. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
8. 12-lead ECG without any clinically significant abnormality as judged by the Investigator, and average QTcB or QTcF < 450 msec or QTc < 480 msec in subjects with Bundle Branch Block.
9. Able to complete all study procedures and planned treatment periods.

Exclusion Criteria:

1. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
2. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
3. Known celiac disease and positive serologic testing for anti-tTG antibodies (required to screen for undiagnosed celiac disease)
4. A positive pre-study drug/alcohol screen.
5. A positive test for HIV antibody.
6. History of regular alcohol consumption within 6 months of the study defined as:

   • an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
7. Unwilling to abstain from alcohol for 48 hours prior to screening, and 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each treatment period.
8. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
9. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
10. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
11. History of sensitivity to the study medication, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
12. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
13. Pregnant females as determined by positive serum hCG test at screening or urine hCG test prior to dosing.
14. Lactating females.
15. The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg, or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects at Screening and pre-dose on Day 1.
16. Unwillingness or inability to follow the procedures outlined in the protocol.
17. Subject is mentally or legally incapacitated.
18. Subject with a medical condition which in the opinion of the investigator and GSK Medical Monitor makes them unsuitable for the study.
19. History of sensitivity to heparin or heparin-induced thrombocytopenia.
20. History of regular use of tobacco- or nicotine-containing products within 6 months prior to screening and unwilling to remain abstinent from tobacco or nicotine containing products for the duration of the study.
21. Consumption of red wine, seville oranges, grapefruit or grapefruit juice, pomegranate, and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-05-05 (Actual); Primary Completion 2010-06-29 (Actual); Study Completion 2010-06-29 (Actual)

PRIMARY OUTCOMES:
Plasma GSK1605786 parameters: AUC(0-∞), AUC(0-t), Cmax. | 2-4 weeks after the last subject last visit

SECONDARY OUTCOMES:
Plasma GSK1605786 parameters: AUC(0-24), %AUCex, tlag, tmax, t1/2 | 2-4 weeks after the last subject last visit
Safety and tolerability parameters including vital signs, ECGs, clinical laboratory | Results will be monitered in real time from screening through to the follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- See also: Results for study 114203 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114203?search=study&study_ids=114203#rs